CLINICAL TRIAL: NCT02224924
Title: Effect of Autologous Blood Patch Injection Versus BioSentry Hydrogel Tract Plug in the Reduction of Pneumothorax Risk Following Lung Biopsy Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-141
Record Dates: First submitted 2014-08-22; First posted 2014-08-25 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-01

CONDITIONS: Lung Biopsy
Keywords: Experimental: autologous blood patch injection (ABPI); Experimental: BioSentry (formerly known as Bio-Seal) hydrogel Tract Plug; 14-141

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- autologous blood patch injection (ABPI) (Active Comparator)
  Interventions: Other: ABPI
- BioSentry (formerly known as Bio-Seal) hydrogel Tract Plug (Experimental)
  Interventions: Device: BioSentry (formerly known as Bio-Seal) hydrogel Tract Plug

INTERVENTIONS:
Other: ABPI — If the patient was assigned to the ABPI group, a blood patch will be administered using the clotted blood in the syringe obtained at the beginning of the procedure. The guiding needle will be retracted up to 1.5-2 cm from the pleural surface, and the blood will be injected steadily and gently as the needle is pulled back out of the pleura. Injection will stop when the operator feels the needle is in subcutaneous tissues.
  Arms: autologous blood patch injection (ABPI)
Device: BioSentry (formerly known as Bio-Seal) hydrogel Tract Plug — If the patient is assigned to BioSentry group, using the manufacturer's deployment device the introducer needle is positioned so that the tip is at least 1.5 cm deep to the visceral pleura. The coaxial introducer needle hub will be prehydrated with a drop of saline, the BioSentry plug housing will be mated and locked to the hub and the plug will be deployed.
  Arms: BioSentry (formerly known as Bio-Seal) hydrogel Tract Plug

SUMMARY:
The purpose of this study is to compare two methods that are currently used at the end of a CT guided lung biopsy to close the hole on the surface of the lung in order to minimize the chance of air leaking out of the hole. The two techniques consist of either injecting a very small amount of your the blood called a blood patch into the biopsy hole or injecting a gel-based FDA approved artificial plug called BioSentry that will eventually get absorbed into the body.

DETAILED DESCRIPTION:
This study will determine the rate of all pneumothoraces and those pneumothoraces requiring treatment following percutaneous lung biopsy in patients who have received ABPI or BioSentry at the end of the biopsy procedure. The data collected will be used to determine if there is equal effectiveness in the reduction of pneumothorax rates from both interventions.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Referred for CT guided biopsy of lung lesion
* Target lesion of any size
* Target lesion located 1.5 cm or more away from visceral pleura based on the needle path
* Skin thickness ≤7 cm (from skin to pleura)
* Needle path without transgression of pleural fissure bleb, or bulla is possible
* Coaxial biopsy technique using Angiotech 19-Gauge introducer needle
* Needle length ≤15

Exclusion Criteria:

* Passage through non-aerated lung or tissue
* More than 1 biopsy on the same side requiring more than 1 pleural puncture
* History of prior ipsilateral lung interventions including:
* Chest tube placement
* Surgery
* Pleurodesis
* Radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2014-08-21 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amgad Moussa, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Maybody M, Muallem N, Brown KT, Moskowitz CS, Hsu M, Zenobi CL, Jihad M, Getrajdman GI, Sofocleous CT, Erinjeri JP, Covey AM, Brody LA, Yarmohammadi H, Deipolyi AR, Bryce Y, Alago W, Siegelbaum RH, Durack JC, Gonzalez-Aguirre AJ, Ziv E, Boas FE, Solomon SB. Autologous Blood Patch Injection versus Hydrogel Plug in CT-guided Lung Biopsy: A Prospective Randomized Trial. Radiology. 2019 Feb;290(2):547-554. doi: 10.1148/radiol.2018181140. Epub 2018 Nov 27. PMID 30480487
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autologous Blood Patch Injection (ABPI) | BioSentry (Formerly Known as Bio-Seal) Hydrogel Tract Plug
Started | 226 | 228
Completed | 156 | 162
Not Completed | 70 | 66
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Biopsy cancelled | 20 | 14
Not completed — Intra procedural exclusion - sealant deployed | 23 | 11
Not completed — Intra procedural exclusion - sealant not deployed | 20 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Blood Patch Injection (ABPI) | BioSentry (Formerly Known as Bio-Seal) Hydrogel Tract Plug | Total
Number analyzed (Participants) | 226 | 227 | 453
Age, Continuous [Mean (Full Range); unit: years] | 66.8 [32 to 92] | 67 [24 to 93] | 67 [24 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 127 | 251
  Male | 102 | 100 | 202
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 21
  Not Hispanic or Latino | 164 | 164 | 328
  Unknown or Not Reported | 51 | 53 | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 10 | 21
  White | 188 | 190 | 378
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 15 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 226 | 227 | 453

OUTCOME MEASURES:

1. Primary Outcome: the Rate of Pneumothorax
Description: within 2 hours following biopsy. Pneumothorax is observed on post procedure CT scan or on follow-up chest radiographs while the patient is in the recovery room, according to standard of care.
Time Frame: 2 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous Blood Patch Injection (ABPI) | BioSentry (Formerly Known as Bio-Seal) Hydrogel Tract Plug
Number analyzed (Participants) | 226 | 228
Participants
  Experienced pneumothorax within 2 hours post procedure | 42 | 60
  Did not experience pneumothorax within 2 hours post procedure | 184 | 168

ADVERSE EVENTS:
Time Frame: 2 weeks post procedure
Arm/Group | Autologous Blood Patch Injection (ABPI) | BioSentry (Formerly Known as Bio-Seal) Hydrogel Tract Plug
All-Cause Mortality (participants affected / at risk) | 0/226 | 0/228
Serious Adverse Events (participants affected / at risk) | 0/226 | 0/228
Other Adverse Events (participants affected / at risk) | 0/226 | 0/228

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT02224924/Prot_SAP_000.pdf